CLINICAL TRIAL: NCT00598312
Title: A Phase 3, Open-Label, Multi-Center, Safety And Efficacy Study of Oakwood Laboratories' Leuprolide Acetate For Injectable Suspension 22.5 mg In Patients With Prostate Cancer
Brief Title: Safety and Efficacy Study of Leuprolide Acetate for Injectable Suspension 22.5 MG in the Treatment of Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oakwood Laboratories, LLC (Industry)
Responsible Party: Edward C. Smith, Chairman, Oakwood Laboratories, LLC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OL-01110
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Leuprolide Acetate for Injectable Suspension — Sustained release injectable microspheres, 22.5 mg, one injection every 84 days, 3-month product

SUMMARY:
The purpose of the study is to demonstrate the safety and efficacy of Leuprolide Acetate for Injectable Suspension 22.5 mg in reducing serum testosterone to castrate levels in patients with prostate cancer.

DETAILED DESCRIPTION:
This study is an open-label, multi-center study in which a minimum of 165 patients will receive one (1) of three (3) lots of Oakwood Laboratories' Leuprolide Acetate for Injectable Suspension 22.5 mg for two cycles. A subset of patients (minimum of 12) will be assigned to each lot (A, B or C) and will have additional blood sampling to characterize leuprolide release kinetics for each dose administered.

ELIGIBILITY:
Inclusion Criteria:

* Reads, understands and is able and willing to sign informed consent form
* Males greater than or equal to age 45
* Histologically and cytologically documented prostate carcinoma
* Candidate for initial hormone therapy - inclusive of patients beginning neoadjuvant or intermittent therapy, being treated locally for advanced disease, or patients beginning therapy for failure of prior local therapy
* Patients who have had prior LHRH therapy in an adjuvant or neoadjuvant setting, providing that the last date of effective therapy was greater than 6 months prior to screening
* ECOG 0-2
* Morning serum testosterone level > 150 ng/dL
* Standard screening labs within 2x ULN (AST, ALT, bilirubin and serum creatinine)
* Hemoglobin > 10 g/dL
* Life expectancy of >1yr.
* Willing to complete both cycles and all procedures of the study

Exclusion Criteria:

* Any prior (except for prior LHRH therapy in an adjuvant or neoadjuvant setting) or current definitive therapy for prostate cancer, including chemotherapy, immunotherapy, tumor-vaccines,biological response modifiers, or estrogens
* Patients who have undergone any prostatic surgery within 4 weeks of Baseline
* Patients who have undergone orchiectomy, adrenalectomy, or hypophysectomy
* Patients that are currently hospitalized or require frequent hospitalization
* Prior resistance to LHRH therapy, either neoadjuvant or adjuvant.
* Patients with evidence of spinal cord compression, ureteral obstruction or clinically significant bladder outlet obstruction
* Participation in any investigational drug, biologic, or device study within five half-lives of its physiological action or three months prior to enrollment, whichever was longer
* Patients anticipated to need concomitant hormonal, anti-androgen, radio-, chemo-, immuno- or surgical therapy for prostate cancer while on study
* History of recent drug and/or alcohol abuse within 6 months of screening
* History of HIV, HCV or HBV infection
* History of hypersensitivity or known allergy to LHRH agonists or antagonists
* Concurrent use of daily corticosteroids or other agents known to modify serum androgen within 12 weeks of screening visit
* Patients on other anti-androgens such as flutamide, nilutamide or bicalutamide
* History of other cancer with the exception of non-metastatic basal or squamous cell carcinoma of the skin
* Patients receiving any type of 5-alpha reductase inhibitor such as Proscar, Propecia, or Avodart within the past 3 months
* Patients who have experienced a myocardial infarction, unstable or uncontrolled cardiovascular disease or a coronary vascular procedure within 6 months of Baseline
* Patients who have experienced venous thrombosis within 6 months of Baseline
* Patients with other serious intercurrent illness(es) or disease(s)that might interfere with, or put them at additional risk for, their ability to receive the treatment outlined in the protocol
* Patients who have a history of the following: Immunization within 4 weeks of Baseline; Flu shots within 2 weeks of Baseline; Donation or receipt of blood or blood products within 2 months of Baseline; Anaphylaxis
* Patients who have received Oakwood's leuprolide acetate formulation previously.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The percentage of responders who attain and maintain castrate levels of serum testosterone | From Day 28 to Day 168.

SECONDARY OUTCOMES:
Safety as shown through laboratory parameters | Day 0 - Day 168
  Hematology, chemistry and urinalysis
Leuprolide serum profiles following administration study drug product. | Day 0 - Day 168
  Leuprolide levels (ng/dL) measured at designated time points to determine a pharmacokinetic profile for the product.
Safety as shown through reported adverse events | Day 0 -168

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Saltzstein, MD, Principal Investigator — Urology San Antonio Research PA; James Page, MD, Study Chair — Oakwood Laboratories, LLC; Beth Glasgow, Study Director — Oakwood Laboratories, LLC
Locations (1):
- Oakwood Laboratories, LLC, Oakwood Village, Ohio, United States